CLINICAL TRIAL: NCT02708160
Title: Assessment of Prevident Sodium Fluoride 1.1% Toothpaste Using an Intra-oral Remineralization-demineralization Model
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn due to business reasons
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ERO-2015-CAI-03-RPS
Record Dates: First submitted 2016-03-04; First posted 2016-03-15 (Estimated); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Tin Fluorides

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fluoride Free toothpaste (Placebo Comparator): Fluoride free (0%), silica based toothpaste
  Interventions: Drug: Fluoride Free toothpaste; Drug: 1.1% Fluoride toothpaste; Drug: 0.243% Fluoride toothpaste
- 1.1% Fluoride toothpaste (Experimental): Prevident 5000 Plus, silica based toothpaste
  Interventions: Drug: Fluoride Free toothpaste; Drug: 1.1% Fluoride toothpaste; Drug: 0.243% Fluoride toothpaste
- 0.243% Fluoride Toothpaste (Active Comparator): silica based fluoride toothpaste
  Interventions: Drug: Fluoride Free toothpaste; Drug: 1.1% Fluoride toothpaste; Drug: 0.243% Fluoride toothpaste

INTERVENTIONS:
Drug: Fluoride Free toothpaste — Brush whole mouth with study toothpaste 2x/day for the 2 week test period. Each brushing routine is 1 minute whole mouth brushing with oral retainer in mouth, spit out toothpaste residue and wait 1 minute before rinsing with water.
  Other Names: Control toothpaste containing no anti-cavity ingredients
Drug: 1.1% Fluoride toothpaste — Brush whole mouth with study toothpaste 2x/day for the 2 week test period. Each brushing routine is 1 minute whole mouth brushing with oral retainer in mouth, spit out toothpaste residue and wait 1 minute before rinsing with water.
  Other Names: Prevident 5000 Plus
Drug: 0.243% Fluoride toothpaste — Brush whole mouth with study toothpaste 2x/day for the 2 week test period. Each brushing routine is 1 minute whole mouth brushing with oral retainer in mouth, spit out toothpaste residue and wait 1 minute before rinsing with water.
  Other Names: silica based fluoride toothpaste

SUMMARY:
This is a double blind, cross-over, controlled clinical trial utilizing thirty (30) adults to evaluate remineralization of early caries lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Male and/or female subjects 18 to 50 years inclusive
2. Minimum of 20 natural uncrowned teeth (excluding third molars) must be present
3. Willing to wear retainer 24 hours per day
4. No active, unrestored cavities
5. Have normal salivary flow rate (stimulated and unstimulated flow of ≥0.7 ml/min and ≥ 0.2 ml/min respectively) ascertained from a preliminary sialometry
6. Available throughout entire study
7. Willing to use only assigned products for oral hygiene throughout the duration of the study
8. Must give written informed consent
9. Must be in good general health
10. No known history of allergy to personal care/consumer products or their ingredients, relevant to any ingredient in the test products as determined by the dental/medical professional monitoring the study

Exclusion Criteria:

1. Advanced periodontal disease
2. Medical condition which requires premedication prior to dental visits/procedures
3. Not enough teeth to secure the oral retainer
4. Diseases of the soft or hard oral tissues
5. Wear an Orthodontic retainer(s)
6. Impaired salivary function
7. Current use drugs that can affect salivary flow
8. Use antibiotics one (1) month prior to or during this study
9. Positive urine test for pregnancy (a urine pregnancy test will be performed on female subjects of child-bearing potential)
10. Participate in another clinical study one (1) week prior to the start of the washout period or during this 9-week study period
11. Use tobacco products
12. Allergic history to common toothpaste ingredients
13. Immune compromised individuals (HIV, AIDS, immuno-suppressive drug therapy) as determined by review of medical history

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Mineral Change (delta Z) | Baseline
  Tooth samples of human enamel are placed in a retainer and worn by each study subject. Enamel block samples will be x-rayed and analyzed for mineral level (volume % of micrometer of lesions, vol % µm) before being placed in the retainer. These baseline values will be compared with the post use delta mineral change ( ΔZ).
Mineral Change (delta Z) | 2 weeks (from Baseline)
  Tooth samples of human enamel are placed in a retainer and worn by each study subject. After 2 weeks of brushing while wearing the study oral retainer, samples from the retainer will be x-rayed and analyzed for mineral level (volume % of micrometer of lesions, vol % µm). These post use values will be compared to the baseline values to give a delta mineral change ( ΔZ).

CONTACTS AND LOCATIONS:
Overall Officials: Bennet Amaechi, PhD, DDS, Principal Investigator — University of Texas

IPD SHARING:
Plan to Share IPD: No